CLINICAL TRIAL: NCT05056181
Title: "MenPhys: Intervention Protocol for Physical Wellness in Mental Health"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Paolo Flocco, adjunct professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 872/CE Lazio 1
Record Dates: First submitted 2021-09-13; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Severe Mental Disorder
MeSH Terms: conditions — Mental Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAI (Experimental): Participants assigned to the PAI arm will receive brief information on the benefits of being more active and will be given information about the best way to training. They will receive conventional medical treatment. They will also participate in 2 weeks of training (12 sessions), plus telematic assistance of a specialized practitioner who will follow them during the post-discharge training sessions for a period of 12 weeks, with 3 workouts per week.
  Interventions: Other: Physical Activity
- TAU (No Intervention): Participants assigned to the TAU arm will receive brief information on the benefits of being more active and will be given information about the best way to training. They will also receive conventional medical treatment.

INTERVENTIONS:
Other: Physical Activity — Physical activity
  Arms: PAI

SUMMARY:
The primary aim of this project is to establish the acceptability of the PAI (physical activity intervention) to service users by evaluating if participants can be recruited into the study and if they complete the intervention.

Secondary aims are to estimate if, compared with treatment as usual (TAU), the PAI intervention (1) positively impacts on subjects' psychiatric symptoms (2) succeeds in improving cardiovascular fitness performance. In addition, will be considered the impact of the PAI versus TAU on sleep behavior, quality of life, drug consumption, reduces sedentary behaviour and unscheduled readmissions to the department within 30 days and within 7 days after their dismission.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any SMI
* Meeting any one of the following criteria as determined by a care co-ordinator:

  1. Overweight
  2. At risk for or have type 2 diabetes mellitus
  3. In the clinician's view, have a sedentary lifestyle
  4. Smoke tobacco
* Ability to provide informed consent
* Ability to understand Italian

Exclusion Criteria:

* under the age of 18
* not having a diagnosis of SMI
* be unable to do exercises
* be unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients that will complete the study (Acceptability) | 24-26 weeks
  to evaluate if participants can be recruited into the study and if they complete the intervention.

SECONDARY OUTCOMES:
Anthropometric measures | 24-26 weeks
  Body Max Index (BMI), in kg/m^2
Anthropometric measures | 24-26 weeks
  height in centimeters
Anthropometric measures | 24-26 weeks
  abdominal circumference in centimeters
Anthropometric measures | 24-26 weeks
  weight in kilograms
Self-report sedentary behaviour and physical activity | 24-26 weeks
  International Physical Activity Questionnaire (IPAQ)
Cardiorespiratory Fitness | 24-26 weeks
  6MWT
Sleep behavior | 24-26 weeks
  Pittsburgh sleep quality index (PSQI)
Quality of life (QoL) | 24-26 weeks
  The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF)
Motivation to engage in physical activity | 24-26 weeks
  Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2)
Psychiatric symptoms | 24-26 weeks
  brief psychiatric rating scale (BPRS)
Psychiatric symptoms | 24-26 weeks
  Hamilton Depression Rating Scale (HAM-D)
Blood samples | 24-26 weeks
  HIgh Density Lipoproteins (HDL)
Blood samples | 24-26 weeks
  blood glucose levels
Blood samples | 24-26 weeks
  insulin levels
Blood samples | 24-26 weeks
  triglycerides
Blood samples | 24-26 weeks
  C-reactive Protein (CRP)
Blood samples | 24-26 weeks
  Low Density Lipoproteins (LDP)